CLINICAL TRIAL: NCT00335816
Title: Timing of Rectal Cancer Response to Chemoradiation
Brief Title: Radiation Therapy and Fluorouracil With or Without Combination Chemotherapy Followed by Surgery in Treating Patients With Stage II or Stage III Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mskcc 12-201; P30CA033572 (NIH); R01CA090559 (NIH); CDR0000458059 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Radiotherapy; Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Closed to Enrollment) (Experimental): All patients undergo chemoradiation therapy comprising radiation therapy once daily 5 days a week for 5 weeks and fluorouracil intravenously continuously over 24 hours 7 days a week for 6 weeks. Patients undergo standard surgical resection after completion of chemoradiation therapy..
  Interventions: Drug: fluorouracil; Procedure: conventional surgery; Radiation: radiation therapy; Other: laboratory biomarker analysis; Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: immunohistochemistry staining method
- Group 2 (Closed to Enrollment) (Experimental): All patients undergo chemoradiation therapy comprising radiation therapy once daily 5 days a week for 5 weeks and fluorouracil IV continuously over 24 hours 7 days a week for 6 weeks. Beginning 4 weeks after completion of chemoradiation therapy, patients receive modified FOLFOX-6 chemotherapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1-2. Treatment repeats every 14 days for 2 courses. After the last week of post-radiation chemotherapy, patients undergo standard surgical resection.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy; Other: laboratory biomarker analysis; Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: immunohistochemistry staining method
- Group 3 (chemotherapy, FOLFOX, conventional surgery) (Experimental): All patients undergo chemoradiation therapy comprising radiation therapy once daily 5 days a week for 5 weeks and fluorouracil IV continuously over 24 hours 7 days a week for 6 weeks. Beginning 4 weeks after completion of chemoradiation therapy, patients receive modified FOLFOX-6 chemotherapy as in group II. Treatment repeats every 14 days for 4 courses. After the last week of post-radiation chemotherapy, patients undergo standard surgical resection.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy; Other: laboratory biomarker analysis; Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: immunohistochemistry staining method
- Group 4 (chemotherapy, FOLFOX, conventional surgery) (Experimental): All patients undergo chemoradiation therapy comprising radiation therapy once daily 5 days a week for 5 weeks and fluorouracil IV continuously over 24 hours 7 days a week for 6 weeks. Beginning 4 weeks after completion of chemoradiation therapy, patients receive modified FOLFOX-6 chemotherapy as in group II. Treatment repeats every 14 days for 6 courses. After the last week of post- radiation chemotherapy, patients undergo standard surgical resection. Patients then receive 3 additional courses of FOLFOX-6 chemotherapy or other chemotherapy off study as directed by the physician.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy; Other: laboratory biomarker analysis; Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: fluorouracil — Given IV
Drug: leucovorin calcium — Given IV
  Arms: Group 2 (Closed to Enrollment); Group 3 (chemotherapy, FOLFOX, conventional surgery); Group 4 (chemotherapy, FOLFOX, conventional surgery)
Drug: oxaliplatin — Given IV
  Arms: Group 2 (Closed to Enrollment); Group 3 (chemotherapy, FOLFOX, conventional surgery); Group 4 (chemotherapy, FOLFOX, conventional surgery)
Procedure: conventional surgery — Patients undergo surgery
Radiation: radiation therapy — Patients undergo radiotherapy
Other: laboratory biomarker analysis — Correlative studies
Genetic: DNA analysis — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as fluorouracil, oxaliplatin, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Fluorouracil may also make tumor cells more sensitive to radiation therapy. Leucovorin calcium may protect normal cells from the side effects of chemotherapy, and it may help fluorouracil work better by making tumor cells more sensitive to the drug. Giving radiation therapy together with chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with fluorouracil with or without combination therapy works in treating patients who are undergoing surgery for stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the rate of pathologic complete response to chemoradiation (no evidence of residual tumor in the resected specimen) of Stage II and Stage III rectal cancers that are staged preoperatively by endorectal ultrasound (ERUS) or magnetic resonance imaging (MRI), treated according to a standardized chemoradiation and surgery protocol, and evaluated by a systematic pathologic exam of the surgical specimen.

II. To study the effect of different chemoradiation-to-surgery intervals on the rate of pathologic complete response, on surgical difficulty, and on postoperative complications.

III. To investigate the feasibility of using sensitive molecular assays to detect tumor cells in the tumor bed and regional lymph nodes of rectal cancer specimens, with or without pathologic complete response to preoperative chemoradiation.

OUTLINE:

Patients are assigned to 1 of 4 treatment groups. All patients undergo chemoradiation therapy comprising radiation therapy once daily 5 days a week for 5 weeks and fluorouracil intravenously (IV) continuously over 24 hours 7 days a week for 6 weeks.

GROUP I (closed to enrollment): Patients undergo standard surgical resection after completion of chemoradiation therapy.

GROUP II (closed to enrollment): Beginning 4 weeks after completion of chemoradiation therapy, patients receive modified FOLFOX-6 chemotherapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1-2. Treatment repeats every 14 days for 2 courses. After the last week of post-radiation chemotherapy, patients undergo standard surgical resection.

GROUP III: Beginning 4 weeks after completion of chemoradiation therapy, patients receive modified FOLFOX-6 chemotherapy as in group II. Treatment repeats every 14 days for 4 courses. After the last week of post-radiation chemotherapy, patients undergo standard surgical resection.

GROUP IV: Beginning 4 weeks after completion of chemoradiation therapy, patients receive modified FOLFOX-6 chemotherapy as in group II. Treatment repeats every 14 days for 6 courses. After the last week of post- radiation chemotherapy, patients undergo standard surgical resection.

In all groups, treatment continues in the absence of disease progression or unacceptable toxicity. A

fter completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an Eastern Cooperative Oncology Group (ECOG) Status of 0 or 1, or comparable Karnofsky performance status
* Patients must have histologically confirmed invasive adenocarcinoma of the rectum Distal border of the tumor must be within 12 cm from the anal verge as measured on rigid proctoscopic exam
* Patients must have Stage II (uT3-4, uN0) or Stage III (any T, uN1-2) tumors, as confirmed by ERUS or MRI; females with anterior tumors invading the posterior vaginal wall (uT4) and males with anterior tumors that invade the seminal vesicles or adjacent organs (uT4) will also be eligible provided they undergo an extended resection including the organs involved
* Patients with high grade obstruction that impedes the ERUS exam are eligible for the study provided they can be staged by MRI
* Patients with synchronous or metachronous colorectal cancer are eligible for the study on condition that they are treated for rectal cancer in accordance with the protocol
* Patients with the following are NOT allowed on study:

  * Metastatic disease or other primaries
  * Locally recurrent rectal cancer
  * Previously documented history of Familial Adenomatous Polyposis
  * History of Inflammatory Bowel Disease
  * History of prior radiation treatments to pelvis
  * History of clinically significant cardiac disease (i.e., Class 3-4 congestive heart failure, symptomatic coronary artery disease, uncontrolled arrhythmia, and/or myocardial infarction within the previous 6 months
  * History of uncontrolled seizures or clinically significant central nervous system disorders
  * History of psychiatric conditions or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance
  * History of allergy and/or hypersensitivity to 5-fluorouracil (fluorouracil), leucovorin (leucovorin calcium), and/or oxaliplatin
  * History of difficulty or inability to take or absorb oral medications
* Patients must have adequate bone marrow, hepatic and renal function within 7 days prior to registration
* White blood cells (WBC) >= 3,000 mm^3
* Absolute neutrophil count (ANC) > 1,500 mm^3
* Hemoglobin > 9.5 mg/dl
* Platelet count >= 100,000 mm^3
* Total bilirubin =< 1.5 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.0 times institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.0 times ULN
* Alkaline phosphatase =< 2.0 times ULN
* Serum creatinine =< 1.5 times ULN
* Patients with hereditary non-polyposis colorectal cancer are eligible for the study provided they meet the rest of the eligibility criteria
* Patients who have experienced a prior malignancy should have received potentially curative therapy for that malignancy, and should be cancer-free for at least five years from the date of initial diagnosis (Exceptions: patients treated for basal cell carcinoma, or carcinoma in-situ of the cervix)
* Patients of reproductive potential should agree to use an effective method of birth control when undergoing treatments with known or possible mutagenic or teratogenic effects; all female participants of childbearing potential must have a negative urine or serum pregnancy test within two weeks prior to study registration
* Patients or the patient's legally acceptable representative must provide written authorization to allow the use and disclosure of protected health information; NOTE: this may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study registration or the initiation of any study-specific procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2008-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of pathologic complete response | Determined at the time of surgery
Effect of different chemoradiation-to-surgery intervals on rate of pathologic complete response and surgical difficulty. | Measured at the time of surgery
Effect of different chemoradiation-to-surgery intervals on postoperative complications | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Julio Garcia-Aguilar, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (15):
- United States (14):
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Medical Center, Duarte, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Colon and Rectal Surgery, Incorporated, Omaha, Nebraska
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
- Tom Baker Cancer Centre - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Pelossof R, Chow OS, Fairchild L, Smith JJ, Setty M, Chen CT, Chen Z, Egawa F, Avila K, Leslie CS, Garcia-Aguilar J. Integrated genomic profiling identifies microRNA-92a regulation of IQGAP2 in locally advanced rectal cancer. Genes Chromosomes Cancer. 2016 Apr;55(4):311-321. doi: 10.1002/gcc.22329. PMID 26865277
- [Derived] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751
- [Derived] Duldulao MP, Lee W, Nelson RA, Li W, Chen Z, Kim J, Garcia-Aguilar J. Mutations in specific codons of the KRAS oncogene are associated with variable resistance to neoadjuvant chemoradiation therapy in patients with rectal adenocarcinoma. Ann Surg Oncol. 2013 Jul;20(7):2166-71. doi: 10.1245/s10434-013-2910-0. Epub 2013 Mar 2. PMID 23456389
- [Derived] Duldulao MP, Lee W, Streja L, Chu P, Li W, Chen Z, Kim J, Garcia-Aguilar J. Distribution of residual cancer cells in the bowel wall after neoadjuvant chemoradiation in patients with rectal cancer. Dis Colon Rectum. 2013 Feb;56(2):142-9. doi: 10.1097/DCR.0b013e31827541e2. PMID 23303141
- [Derived] Duldulao MP, Lee W, Nelson RA, Ho J, Le M, Chen Z, Li W, Kim J, Garcia-Aguilar J. Gene polymorphisms predict toxicity to neoadjuvant therapy in patients with rectal cancer. Cancer. 2013 Mar 1;119(5):1106-12. doi: 10.1002/cncr.27862. Epub 2012 Oct 23. PMID 23096768
- [Derived] Chen Z, Liu Z, Deng X, Warden C, Li W, Garcia-Aguilar J. Chromosomal copy number alterations are associated with persistent lymph node metastasis after chemoradiation in locally advanced rectal cancer. Dis Colon Rectum. 2012 Jun;55(6):677-85. doi: 10.1097/DCR.0b013e31824f873f. PMID 22595848
- [Derived] Duldulao MP, Lee W, Le M, Wiatrek R, Nelson RA, Chen Z, Li W, Kim J, Garcia-Aguilar J. Surgical complications and pathologic complete response after neoadjuvant chemoradiation in locally advanced rectal cancer. Am Surg. 2011 Oct;77(10):1281-5. PMID 22127070
- [Derived] Garcia-Aguilar J, Chen Z, Smith DD, Li W, Madoff RD, Cataldo P, Marcet J, Pastor C. Identification of a biomarker profile associated with resistance to neoadjuvant chemoradiation therapy in rectal cancer. Ann Surg. 2011 Sep;254(3):486-92; discussion 492-3. doi: 10.1097/SLA.0b013e31822b8cfa. PMID 21865946
- [Derived] Duldulao MP, Lee W, Le M, Chen Z, Li W, Wang J, Gao H, Li H, Kim J, Garcia-Aguilar J. Gene expression variations in microsatellite stable and unstable colon cancer cells. J Surg Res. 2012 May 1;174(1):1-6. doi: 10.1016/j.jss.2011.06.016. Epub 2011 Jul 7. PMID 21816436
- [Derived] Chen Z, Liu Z, Li W, Qu K, Deng X, Varma MG, Fichera A, Pigazzi A, Garcia-Aguilar J. Chromosomal copy number alterations are associated with tumor response to chemoradiation in locally advanced rectal cancer. Genes Chromosomes Cancer. 2011 Sep;50(9):689-99. doi: 10.1002/gcc.20891. Epub 2011 May 16. PMID 21584903
- [Derived] Garcia-Aguilar J, Smith DD, Avila K, Bergsland EK, Chu P, Krieg RM; Timing of Rectal Cancer Response to Chemoradiation Consortium. Optimal timing of surgery after chemoradiation for advanced rectal cancer: preliminary results of a multicenter, nonrandomized phase II prospective trial. Ann Surg. 2011 Jul;254(1):97-102. doi: 10.1097/SLA.0b013e3182196e1f. PMID 21494121
- [Derived] Chen Z, Duldulao MP, Li W, Lee W, Kim J, Garcia-Aguilar J. Molecular diagnosis of response to neoadjuvant chemoradiation therapy in patients with locally advanced rectal cancer. J Am Coll Surg. 2011 Jun;212(6):1008-1017.e1. doi: 10.1016/j.jamcollsurg.2011.02.024. Epub 2011 Mar 31. PMID 21458303
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/